CLINICAL TRIAL: NCT02517580
Title: Vitamin K2 Supplementation and Effect on Arterial Stiffness Progression in the Renal Transplant Population
Brief Title: Vitamin K2 Supplementation and Arterial Stiffness in the Renal Transplant Population (The KING Trial)
Acronym: KING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lebanese American University (Other)
Collaborators: Omicron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sola Aoun Bahous, M.D. Ph.D., Associate Professor of Medicine, Division of Nephrology and Transplantation, Lebanese American University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK7-002
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-08

CONDITIONS: Arterial Stiffness; Vitamin K2 Deficiency
MeSH Terms: interventions — Vitamin K 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin K2 (MK7) (Experimental): Vitamin K2 (MK7) 360 mcg/day PO once daily for 8 weeks
  Interventions: Dietary Supplement: Vitamin K2 (MK7)

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (MK7)
  Other Names: MenaQ7

SUMMARY:
This study is a single arm, single center clinical trial that aims to evaluate the effect of 8 weeks of vitamin K2 replacement (360 mcg/day) on the progression of arterial stiffness in stable renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Functional renal graft
* Stable renal function for at least 3 months prior to enrollment

Exclusion Criteria:

* History of thrombotic events
* Diagnosed coagulopathy
* Cardiovascular event in the past month prior to enrollment
* Current or planned pregnancy
* Lactation
* Soy allergy
* Concomitant or recent (past 6 months) use of supplements that contain vitamin K
* Warfarin treatment
* Known intestinal malabsorption or hypomotility syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sola Aoun Bahous, M.D. Ph.D., Principal Investigator — Lebanese American University
Locations (1):
- Lebanese American University Medical Center - Rizk Hospital, El Achrafiyé, Beyrouth, Lebanon

REFERENCES:
- [Background] Mansour AG, Hariri E, Daaboul Y, Korjian S, El Alam A, Protogerou AD, Kilany H, Karam A, Stephan A, Bahous SA. Vitamin K2 supplementation and arterial stiffness among renal transplant recipients-a single-arm, single-center clinical trial. J Am Soc Hypertens. 2017 Sep;11(9):589-597. doi: 10.1016/j.jash.2017.07.001. Epub 2017 Jul 13. PMID 28756183

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin K2 (MK7)
Started | 60
Completed | 56
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin K2 (MK7)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Lebanon | 60
Transplantation duration [Mean (Standard Deviation); unit: years] | 15.9 (6)

OUTCOME MEASURES:

1. Primary Outcome: Reduction From Baseline in Carotid-femoral Pulse Wave Velocity at 8 Weeks
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: m/s
Groups:
- Vitamin K2 (MK7): Vitamin K2 (MK7) 360 mcg/day PO once daily for 8 weeks
  Vitamin K2 (MK7)
Arm/Group | Vitamin K2 (MK7)
Number analyzed (Participants) | 56
m/s | -1.4 (0.2)

2. Secondary Outcome: Change From Baseline in Central Pressure by Ambulatory Hemodynamic Measurement (Mobil-O-Graph) at 8 Weeks
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Augmentation Index by Ambulatory Hemodynamic Measurement (Mobil-O-Graph) at 8 Weeks
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Blood Concentration of Dephosphorylated-uncarboxylated Matrix Gla Protein (Dp-ucMGP) at 8 Weeks
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Vitamin K2 (MK7)
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 12/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin K2 (MK7) (N=60)
GI symptoms (Gastrointestinal disorders) | 9 (60)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (60)
Acute kidney injury (Renal and urinary disorders) | 2 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No